CLINICAL TRIAL: NCT00672659
Title: Phase IIa Proof of Concept Study of Pipamperone/Citalopram (PipCit) Versus Citalopram in the Treatment of Major Depressive Disorder (MDD)
Brief Title: Pipamperone/Citalopram (PipCit)Versus Citalopram in the Treatment of Major Depressive Disorder(MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaNeuroBoost N.V. (Industry)
Responsible Party: Erik Buntinx, MD, PharmaNeuroBoost N.V.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PNB/CPS 02 2007
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Depression
Keywords: Lost of interest, Depressed Mood
MeSH Terms: conditions — Depression; Consciousness Disorders | interventions — Citalopram; pipamperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Citalopram, 40 mg daily in combination with Pipamperone, 5 mg twice daily (bd)
  Interventions: Drug: Citalopram + Pipamperone
- 2 (Placebo Comparator): Citalopram, 40 mg daily in combination with Placebo, dummy twice daily (bd)
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram + Pipamperone — Citalopram, 40 mg daily, 8 weeks Pipamperone, 5 mg twice daily, 8 weeks
  Arms: 1
Drug: Citalopram — Citalopram, 40 mg daily, 8 weeks Placebo, dummy, twice a day, 8 weeks
  Arms: 2

SUMMARY:
The primary objective is to demonstrate whether the addition of pipamperone 5 mg twice daily (bd) to citalopram, 40 mg daily in patients suffering from MDD will improve the efficacy of citalopram 40 mg in these patients.

Secondary objectives are to demonstrate whether the addition of pipamperone 5 mg twice daily (bd) to citalopram, 40 mg daily in patients suffering from MDD:

1. Will increase the rate of resolution of symptoms with citalopram 40 mg.
2. Show the combined product to be safe and tolerable.

Patients are scheduled to receive study medication for eight weeks and a final follow-up check will be carried out 28 days after completing the study.

All patients will receive active citalopram from baseline and will be randomised to receive either active pipamperone or a placebo equivalent for eight weeks during which time they will attend for 6 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* 18-65 years inclusive
* Suffering from a moderate to severe MDD as defined by DSM IV with an existence of depressed mood and loss of interest/anhedonia for at least four weeks and no longer than six months for the current episode
* Diagnosis will be confirmed by the Mini International Neuropsychiatric Interview (MINI) version 5.0.0.
* Clinical global impression - severity scale (CGI-S) rating of at least four and a minimum Hamilton Depression Scale (HAM-D) 17 items total score of 18 at screen and baseline
* A non-psychotic state
* Where appropriate, male patients should agree to use barrier contraceptive measures (condoms) during the course of the study and for three months after the last dose of medication

Exclusion Criteria:

* Premenopausal females not using adequate contraceptive measures
* Considered by the investigator to be a significant risk of suicide or scoring 5 or more on the MADRS question 10
* Significant other psychiatric illness which would interfere with trial assessments - co-morbid generalised anxiety disorder (GAD) and panic disorder will be permitted where MDD is considered the primary diagnosis
* Significant physical illness which would interfere with trial assessments
* Reduced hepatic function
* Epilepsy
* History of cardiac dysrhythmia
* Alcohol intake above accepted UK ranges
* Recent (1 week) antidepressant (except for fluoxetine - 4 weeks and St John's Wort or MAOI's - 14 days), benzodiazepine or any other psychotropic medication ingestion including lithium or other mood stabilisers
* Resistant depression defined as having failed to respond to

  * Two previous antidepressants at an adequate dose ingested for at least 4 weeks during the current episode
  * To an augmentation therapy with an atypical antipsychotic drug
* Electroconvulsive therapy (ECT) for the current episode
* Formal psychotherapy or alternative treatments for one week prior to or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale score | 8 weeks

SECONDARY OUTCOMES:
The number of patients showing evidence of onset of action defined as a 20% improvement from baseline MADRS | At Weeks 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Erik Buntinx, MD, Study Chair — PharmaNeuroBoost N.V.; Alan Wade, MG, Study Director — CPSResearch; Gordon Crawford, MD, Principal Investigator — CPSResearch
Locations (1):
- CPSResearch, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] Wade AG, Crawford GM, Nemeroff CB, Schatzberg AF, Schlaepfer T, McConnachie A, Haazen L, Buntinx E. Citalopram plus low-dose pipamperone versus citalopram plus placebo in patients with major depressive disorder: an 8-week, double-blind, randomized study on magnitude and timing of clinical response. Psychol Med. 2011 Oct;41(10):2089-97. doi: 10.1017/S0033291711000158. Epub 2011 Feb 25. PMID 21349239
- See also: Pubmed abstract — http://www.ncbi.nlm.nih.gov/pubmed/21349239